CLINICAL TRIAL: NCT04272112
Title: Clinical Performance of All-ceramic Posterior Crowns. A Randomized, Prospective Clinical Trial Comparing Glass-ceramic Crowns to Monolithic Translucent Zirconia Crowns With and Without a Semi-veneer
Brief Title: Clinical Performance of All-ceramic Posterior Crowns. A Randomized, Prospective Clinical.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Minh Le, Prinicipal investigator, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN1401
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Dental Prosthesis Failure
Keywords: all ceramic; zirconia; crown; clinal trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glass-ceramic (Active Comparator): 30 dental crowns of lithium-disilicate glass-ceramic
  Interventions: Combination Product: BruxZir, Glidewell; Combination Product: BruxZir*, Glidewell
- Zirconia (Active Comparator): 30 dental crowns of high translucent zirconia
  Interventions: Combination Product: IPS e.max CAD, Ivoclar Vivadent; Combination Product: BruxZir*, Glidewell
- Zirconia with mini-veneer (Active Comparator): 30 dental crowns of high translucent zirconia with a mini-veneer of porcelain
  Interventions: Combination Product: IPS e.max CAD, Ivoclar Vivadent; Combination Product: BruxZir, Glidewell

INTERVENTIONS:
Combination Product: IPS e.max CAD, Ivoclar Vivadent — Type: monolithic lithium-disilicate glass ceramic
  Arms: Zirconia; Zirconia with mini-veneer
Combination Product: BruxZir, Glidewell — Type: high translucent zirconia
  Arms: Glass-ceramic; Zirconia with mini-veneer
Combination Product: BruxZir*, Glidewell — Type: high translucent zirconia with a mini-veneer of porcelain
  Arms: Glass-ceramic; Zirconia

SUMMARY:
This is a randomized, prospective clinical trial. The aim of the project is to assess the clinical performance of three types of tooth-supported crowns; monolithic high translucent colored zirconia, crowns of high-translucent colored zirconia with a mini-veneer buccally and crowns of lithium-disilicate glass-ceramic. Crowns will be placed on posterior teeth and evaluated from an esthetic and functional point of view, to identify if there are any differences between the materials.

DETAILED DESCRIPTION:
90 monolithic tooth-supported crowns are planned to be included in the study; 30 crowns of high translucent zirconia (BruxZir, Glidewell), 30 crowns of high translucent zirconia (BruxZir, Glidewell) with a mini-veneer of porcelain and 30 crowns of lithium-disilicate glass-ceramic (IPS e.max CAD, Ivoclar Vivadent AG, Schaan, Liechtenstein).

Patients with indications for single crowns will be recruited from three general dental clinics. Inclusion criteria for participating in this study are patients in need of crowns in the posterior dentition, premolars and molars. Exclusion criteria are patients with high caries activity/risk for caries and/or advanced periodontal disease. Patients who meet the criteria will be offered the opportunity to participate in the study. They will receive written information about the study design, clinical procedures and the materials and methods to be used. Patients who are interested will confirm their participation by a written consent. The patients will be offered an extended warranty for the crowns in case of failure.

The study has been approved by the Regional Ethical Board in Lund, Sweden

ELIGIBILITY:
Inclusion criteria:

* need of one or more dental crowns in the posterior dentition, premolars and molars

Exclusion criteria:

* high caries activity/risk for caries and/or advanced periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical perfomance | 12 month
  To identify if there are any differences between the materials. The marginal integrity and surface will be rated as excellent, acceptable, retrievable or not acceptable according to a modified California Dental Association (CDA) quality assessment system.
Clinical perfomance | 24 month
  To identify if there are any differences between the materials. The marginal integrity and surface will be rated as excellent, acceptable, retrievable or not acceptable according to a modified California Dental Association (CDA) quality assessment system.
Clinical perfomance | 36 month
  To identify if there are any differences between the materials. The marginal integrity and surface will be rated as excellent, acceptable, retrievable or not acceptable according to a modified California Dental Association (CDA) quality assessment system.
Clinical perfomance | 60 month
  To identify if there are any differences between the materials. The marginal integrity and surface will be rated as excellent, acceptable, retrievable or not acceptable according to a modified California Dental Association (CDA) quality assessment system.

SECONDARY OUTCOMES:
Patient questionnaire | 12 month
  Self-reported satisfaction with their treatment from 0 ('not satisfied at all') to 10 ('completely satisfied').
Patient questionnaire | 24 month
  Self-reported satisfaction with their treatment from 0 ('not satisfied at all') to 10 ('completely satisfied').
Patient questionnaire | 36 month
  Self-reported satisfaction with their treatment from 0 ('not satisfied at all') to 10 ('completely satisfied').
Patient questionnaire | 60 month
  Self-reported satisfaction with their treatment from 0 ('not satisfied at all') to 10 ('completely satisfied').

CONTACTS AND LOCATIONS:
Overall Officials: Christel Larsson, PhD, Study Chair — Malmö University
Locations (1):
- Malmö University, Malmo, Sweden

REFERENCES:
- [Background] Le M, Papia E, Larsson C. The clinical success of tooth- and implant-supported zirconia-based fixed dental prostheses. A systematic review. J Oral Rehabil. 2015 Jun;42(6):467-80. doi: 10.1111/joor.12272. Epub 2015 Jan 10. PMID 25580846
- [Background] LE M, Larsson C, Papia E. Bond strength between MDP-based cement and translucent zirconia. Dent Mater J. 2019 Jun 1;38(3):480-489. doi: 10.4012/dmj.2018-194. Epub 2019 May 17. PMID 31105161
- [Background] Larsson C, Wennerberg A. The clinical success of zirconia-based crowns: a systematic review. Int J Prosthodont. 2014 Jan-Feb;27(1):33-43. doi: 10.11607/ijp.3647. PMID 24392475
- [Background] Johansson C, Kmet G, Rivera J, Larsson C, Vult Von Steyern P. Fracture strength of monolithic all-ceramic crowns made of high translucent yttrium oxide-stabilized zirconium dioxide compared to porcelain-veneered crowns and lithium disilicate crowns. Acta Odontol Scand. 2014 Feb;72(2):145-53. doi: 10.3109/00016357.2013.822098. Epub 2013 Jul 18. PMID 23865549